CLINICAL TRIAL: NCT02069418
Title: Could Positon Emission Tomography With Radiolabelled 3'-Deoxy-3'-(18)F-Fluoro-L-Thymidine be a Theranostic Tool During Erlotinib Treatment in Non-small Cell Lung Cancer Patients ?
Brief Title: Theranostic Tool During Erlotinib Treatment in Non-small Cell Lung Cancer Patient
Acronym: FLT-THERA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: University Hospital, Tours (Other); Army Hospital, Percy (Unknown); Créteil Hospital (Other); University Hospital, Rouen (Other); Central Hospital, Nancy, France (Other); University Hospital, Toulouse (Other); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PHRC 2012-01; 2013-001301-87 (EudraCT Number)
Record Dates: First submitted 2014-02-12; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Non-small Cell Lung Cancer Metastatic or Non-small Cell Lung Cancer Recurrent; No EGFR Activating Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental): All patients will be in the same arm. Patients are going to have two 18F-FLT-TEP and two 18F-FDG-TEP : the first ones during the two weeks before the beginning of erlotinib and the second ones will occur during the second week after the initiation of erlotinib. The order of TEP is not definite : 18F-FLT-TEP may be planned first or reciprocally. A period of 48 hours must separate two TEP.
  Interventions: Radiation: 18F-FLT-TEP; Radiation: 18F-FDG-TEP

INTERVENTIONS:
Radiation: 18F-FLT-TEP — Patients are going to have two 18F-FLT-TEP : one during the two weeks before the beginning of erlotinib and the second one will occur during the second week after the initiation of erlotinib.
Radiation: 18F-FDG-TEP — Patients are going to have two 18F-FDG-TEP : one during the two weeks before the beginning of erlotinib and the second one will occur during the second week after the initiation of erlotinib.

SUMMARY:
In France, lung cancer is the leading cause of death induced by cancer. Therapeutic advances have been made in therapy of unresectable non-small cell lung cancer (NSCLC) with tyrosine kinase receptor inhibitors blocking the Epidermal Growth Factor Receptor (EGFR), as erlotinib.

This drug usually does not induce rapid shrinking of NSCLC tumour explaining why RECIST criteria are less reliable with erlotinib than cytotoxic drugs after 8 weeks of treatment.

Among patients with unresectable NSCLC, 3'-deoxy-3'-18F-fluoro-L-thymidine (18F-FLT) and 18F-2-18F-fluoro-2-deoxy-D-glucose (18F- FDG) Positron Emission Tomography (PET) has identified early responding patients and with better progression-free survival in erlotinib first line and in the second or third line.

To date, none medico-economic study has been conducted to determine if this strategy will be cost-effective.

The purpose of this study is to confirm that an early metabolic imaging with 18 F-FLT and 18FFDG PET could have theranostic issue by identifying at the fourteenth day of erlotinib (second line or more) the subjects that do not respond to erlotinib, i.e. 6 weeks prior to the morphological evaluation based on the new RECIST 1.1, that is typically done at week 8 of erlotinib treatment.

A health economics ancillary study will be achieved. Indeed, recent therapeutic improvements, in particular targeted therapies in NSCLC, have improved quality of life and life expectancy, but have also induce an important increase of the health costs. According to studies, the mean cost of the treatments of NSCLC has been increased by a factor 3 during the 10 last years. More efficient strategies that would permit to stop early with objective endpoints, expensive therapies is a main achievement in thoracic oncology.

The potential clinical impacts of this work are 1) to stop early erlotinib in non-responders and replace another treatment before a deterioration in their physical status, 2) reduce the risk of side effects and costs of unnecessary treatment and 3) to propose a customization treatment after the first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* age over superior to 18
* NSCLC proved by a histological biopsy
* EGFR mutation status known with no activating EGFR mutation
* indication of erlotinib therapy after at least one previous therapy
* patients who have signed an informed consent to participate in this study
* life expectancy exceeding 12 weeks
* WHO activity score between 0 and 2.

Exclusion Criteria:

* contraindication for the initiation of erlotinib
* refusal to sign the consent
* progressive inflammatory disease
* infection with the HIV virus
* other malignant disease
* life expectancy less than 12 weeks
* major adults protected by French law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Early prediction of response to erlotinib therapy by 18F-FLT and 18F-FDG PETscans | Six months
  The primary endpoint is the correlation between tumour response to erlotinib assessed by morphological imaging by RECIST 1.1 at Day 56 (considered the gold standard) and the change in the uptake of 18F-FLT and 18F-FDG assessed by PET before and at Day 7 after initiation of erlotinib derived from criteria PERCIST. the Kappa test will be used.

SECONDARY OUTCOMES:
Economic study of the early prediction of response to erlotinib therapy by 18F-FLT and 18F-FDG PETscans | Six months
  The aim of this study will be to determine if health costs could be minimized by early prediction of response to erltinib therapy.

CONTACTS AND LOCATIONS:
Overall Officials: José HUREAUX, MD, PhD, Principal Investigator — University Hospital, Angers; Olivier COUTURIER, MD, PhD, Study Chair — University Hospital, Angers
Locations (8):
- France (8):
  - University Hospital, Bordeaux, Bordeaux, Gironde
  - Army Hospital, Percy, Percy, Haut de Seine
  - University Hospital, Toulouse, Toulouse, Haute Garonne
  - University Hospital, Tours, Tours, Indre et Loire
  - University Hospital, Angers, Angers, Maine et Loire
  - University Hospital, Nancy, Nancy, Meurthe et Moselle
  - University Hospital, Rouen, Rouen, Seine maritime
  - Hospital, Créteil, Créteil, Val de Marne

REFERENCES:
- [Background] Vesselle H, Grierson J, Muzi M, Pugsley JM, Schmidt RA, Rabinowitz P, Peterson LM, Vallieres E, Wood DE. In vivo validation of 3'deoxy-3'-[(18)F]fluorothymidine ([(18)F]FLT) as a proliferation imaging tracer in humans: correlation of [(18)F]FLT uptake by positron emission tomography with Ki-67 immunohistochemistry and flow cytometry in human lung tumors. Clin Cancer Res. 2002 Nov;8(11):3315-23. PMID 12429617
- [Background] Aouba A, Pequignot F, Le Toullec A, Jougla E. Les causes médicales de décès en France en 2004 et leur évolution 1980-2004. Bul Epidémiol Hebd 2007;35-36:308-14.
- [Background] Ferlay J, Parkin DM, Steliarova-Foucher E. Estimates of cancer incidence and mortality in Europe in 2008. Eur J Cancer. 2010 Mar;46(4):765-81. doi: 10.1016/j.ejca.2009.12.014. Epub 2010 Jan 29. PMID 20116997
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol 2012;13:239-46.
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Chouaid C, Moser A, Coudray-Omnes C, Vergnenegre A. [Economic impact of second- and third-line erlotinib treatment of non small-cell lung cancer]. Rev Mal Respir. 2008 Nov;25(9):1096-103. doi: 10.1016/s0761-8425(08)74979-9. French. PMID 19106905
- [Background] Miller AB, Hoogstraten B, Staquet M, Winkler A. Reporting results of cancer treatment. Cancer. 1981 Jan 1;47(1):207-14. doi: 10.1002/1097-0142(19810101)47:13.0.co;2-6. PMID 7459811
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Shankar LK, Hoffman JM, Bacharach S, Graham MM, Karp J, Lammertsma AA, Larson S, Mankoff DA, Siegel BA, Van den Abbeele A, Yap J, Sullivan D; National Cancer Institute. Consensus recommendations for the use of 18F-FDG PET as an indicator of therapeutic response in patients in National Cancer Institute Trials. J Nucl Med. 2006 Jun;47(6):1059-66. No abstract available. PMID 16741317
- [Background] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Background] Dittmann H, Dohmen BM, Kehlbach R, Bartusek G, Pritzkow M, Sarbia M, Bares R. Early changes in [18F]FLT uptake after chemotherapy: an experimental study. Eur J Nucl Med Mol Imaging. 2002 Nov;29(11):1462-9. doi: 10.1007/s00259-002-0925-z. Epub 2002 Sep 6. PMID 12397465
- [Background] Barthel H, Perumal M, Latigo J, He Q, Brady F, Luthra SK, Price PM, Aboagye EO. The uptake of 3'-deoxy-3'-[18F]fluorothymidine into L5178Y tumours in vivo is dependent on thymidine kinase 1 protein levels. Eur J Nucl Med Mol Imaging. 2005 Mar;32(3):257-63. doi: 10.1007/s00259-004-1611-0. Epub 2004 Sep 4. PMID 15791434
- [Background] Oyama N, Ponde DE, Dence C, Kim J, Tai YC, Welch MJ. Monitoring of therapy in androgen-dependent prostate tumor model by measuring tumor proliferation. J Nucl Med. 2004 Mar;45(3):519-25. PMID 15001697
- [Background] Sugiyama M, Sakahara H, Sato K, Harada N, Fukumoto D, Kakiuchi T, Hirano T, Kohno E, Tsukada H. Evaluation of 3'-deoxy-3'-18F-fluorothymidine for monitoring tumor response to radiotherapy and photodynamic therapy in mice. J Nucl Med. 2004 Oct;45(10):1754-8. PMID 15471845
- [Background] Graf N, Herrmann K, den Hollander J, Fend F, Schuster T, Wester HJ, Senekowitsch-Schmidtke R, zum Buschenfelde CM, Peschel C, Schwaiger M, Dechow T, Buck AK. Imaging proliferation to monitor early response of lymphoma to cytotoxic treatment. Mol Imaging Biol. 2008 Nov-Dec;10(6):349-55. doi: 10.1007/s11307-008-0162-3. Epub 2008 Aug 14. PMID 18704591
- [Background] Jensen MM, Erichsen KD, Bjorkling F, Madsen J, Jensen PB, Hojgaard L, Sehested M, Kjaer A. Early detection of response to experimental chemotherapeutic Top216 with [18F]FLT and [18F]FDG PET in human ovary cancer xenografts in mice. PLoS One. 2010 Sep 24;5(9):e12965. doi: 10.1371/journal.pone.0012965. PMID 20885974
- [Background] Leyton J, Latigo JR, Perumal M, Dhaliwal H, He Q, Aboagye EO. Early detection of tumor response to chemotherapy by 3'-deoxy-3'-[18F]fluorothymidine positron emission tomography: the effect of cisplatin on a fibrosarcoma tumor model in vivo. Cancer Res. 2005 May 15;65(10):4202-10. doi: 10.1158/0008-5472.CAN-04-4008. PMID 15899811
- [Background] Apisarnthanarax S, Alauddin MM, Mourtada F, Ariga H, Raju U, Mawlawi O, Han D, Bornmann WG, Ajani JA, Milas L, Gelovani JG, Chao KS. Early detection of chemoradioresponse in esophageal carcinoma by 3'-deoxy-3'-3H-fluorothymidine using preclinical tumor models. Clin Cancer Res. 2006 Aug 1;12(15):4590-7. doi: 10.1158/1078-0432.CCR-05-2720. PMID 16899606
- [Background] Molthoff CF, Klabbers BM, Berkhof J, Felten JT, van Gelder M, Windhorst AD, Slotman BJ, Lammertsma AA. Monitoring response to radiotherapy in human squamous cell cancer bearing nude mice: comparison of 2'-deoxy-2'-[18F]fluoro-D-glucose (FDG) and 3'-[18F]fluoro-3'-deoxythymidine (FLT). Mol Imaging Biol. 2007 Nov-Dec;9(6):340-7. doi: 10.1007/s11307-007-0104-5. PMID 17643202
- [Background] Atkinson DM, Clarke MJ, Mladek AC, Carlson BL, Trump DP, Jacobson MS, Kemp BJ, Lowe VJ, Sarkaria JN. Using fluorodeoxythymidine to monitor anti-EGFR inhibitor therapy in squamous cell carcinoma xenografts. Head Neck. 2008 Jun;30(6):790-9. doi: 10.1002/hed.20770. PMID 18286491
- [Background] Ullrich RT, Zander T, Neumaier B, Koker M, Shimamura T, Waerzeggers Y, Borgman CL, Tawadros S, Li H, Sos ML, Backes H, Shapiro GI, Wolf J, Jacobs AH, Thomas RK, Winkeler A. Early detection of erlotinib treatment response in NSCLC by 3'-deoxy-3'-[F]-fluoro-L-thymidine ([F]FLT) positron emission tomography (PET). PLoS One. 2008;3(12):e3908. doi: 10.1371/journal.pone.0003908. Epub 2008 Dec 12. PMID 19079597
- [Background] Wei LH, Su H, Hildebrandt IJ, Phelps ME, Czernin J, Weber WA. Changes in tumor metabolism as readout for Mammalian target of rapamycin kinase inhibition by rapamycin in glioblastoma. Clin Cancer Res. 2008 Jun 1;14(11):3416-26. doi: 10.1158/1078-0432.CCR-07-1824. PMID 18519772
- [Background] Brepoels L, Stroobants S, Verhoef G, De Groot T, Mortelmans L, De Wolf-Peeters C. (18)F-FDG and (18)F-FLT uptake early after cyclophosphamide and mTOR inhibition in an experimental lymphoma model. J Nucl Med. 2009 Jul;50(7):1102-9. doi: 10.2967/jnumed.109.062208. Epub 2009 Jun 12. PMID 19525456
- [Background] Buck AK, Kratochwil C, Glatting G, Juweid M, Bommer M, Tepsic D, Vogg AT, Mattfeldt T, Neumaier B, Moller P, Reske SN. Early assessment of therapy response in malignant lymphoma with the thymidine analogue [18F]FLT. Eur J Nucl Med Mol Imaging. 2007 Nov;34(11):1775-82. doi: 10.1007/s00259-007-0452-z. Epub 2007 May 31. PMID 17541585
- [Background] McKinley ET, Ayers GD, Smith RA, Saleh SA, Zhao P, Washington MK, Coffey RJ, Manning HC. Limits of [18F]-FLT PET as a biomarker of proliferation in oncology. PLoS One. 2013;8(3):e58938. doi: 10.1371/journal.pone.0058938. Epub 2013 Mar 15. PMID 23554961
- [Background] Lawrence J, Vanderhoek M, Barbee D, Jeraj R, Tumas DB, Vail DM. Use of 3'-deoxy-3'-[18F]fluorothymidine PET/CT for evaluating response to cytotoxic chemotherapy in dogs with non-Hodgkin's lymphoma. Vet Radiol Ultrasound. 2009 Nov-Dec;50(6):660-8. doi: 10.1111/j.1740-8261.2009.01612.x. PMID 19999354
- [Background] Sohn HJ, Yang YJ, Ryu JS, Oh SJ, Im KC, Moon DH, Lee DH, Suh C, Lee JS, Kim SW. [18F]Fluorothymidine positron emission tomography before and 7 days after gefitinib treatment predicts response in patients with advanced adenocarcinoma of the lung. Clin Cancer Res. 2008 Nov 15;14(22):7423-9. doi: 10.1158/1078-0432.CCR-08-0312. PMID 19010859
- [Background] Zander T, Scheffler M, Nogova L, Kobe C, Engel-Riedel W, Hellmich M, Papachristou I, Toepelt K, Draube A, Heukamp L, Buettner R, Ko YD, Ullrich RT, Smit E, Boellaard R, Lammertsma AA, Hallek M, Jacobs AH, Schlesinger A, Schulte K, Querings S, Stoelben E, Neumaier B, Thomas RK, Dietlein M, Wolf J. Early prediction of nonprogression in advanced non-small-cell lung cancer treated with erlotinib by using [(18)F]fluorodeoxyglucose and [(18)F]fluorothymidine positron emission tomography. J Clin Oncol. 2011 May 1;29(13):1701-8. doi: 10.1200/JCO.2010.32.4939. Epub 2011 Mar 21. PMID 21422426
- [Background] Mileshkin L, Hicks RJ, Hughes BG, Mitchell PL, Charu V, Gitlitz BJ, Macfarlane D, Solomon B, Amler LC, Yu W, Pirzkall A, Fine BM. Changes in 18F-fluorodeoxyglucose and 18F-fluorodeoxythymidine positron emission tomography imaging in patients with non-small cell lung cancer treated with erlotinib. Clin Cancer Res. 2011 May 15;17(10):3304-15. doi: 10.1158/1078-0432.CCR-10-2763. Epub 2011 Mar 1. PMID 21364032
- [Background] Benz MR, Herrmann K, Walter F, Garon EB, Reckamp KL, Figlin R, Phelps ME, Weber WA, Czernin J, Allen-Auerbach MS. (18)F-FDG PET/CT for monitoring treatment responses to the epidermal growth factor receptor inhibitor erlotinib. J Nucl Med. 2011 Nov;52(11):1684-1689. doi: 10.2967/jnumed.111.095257. PMID 22045706
- [Background] Girard N, Sima CS, Jackman DM, Sequist LV, Chen H, Yang JC, Ji H, Waltman B, Rosell R, Taron M, Zakowski MF, Ladanyi M, Riely G, Pao W. Nomogram to predict the presence of EGFR activating mutation in lung adenocarcinoma. Eur Respir J. 2012 Feb;39(2):366-72. doi: 10.1183/09031936.00010111. Epub 2011 Jul 20. PMID 21778168
- [Background] Garassino MC, Martelli O, Broggini M, Farina G, Veronese S, Rulli E, Bianchi F, Bettini A, Longo F, Moscetti L, Tomirotti M, Marabese M, Ganzinelli M, Lauricella C, Labianca R, Floriani I, Giaccone G, Torri V, Scanni A, Marsoni S; TAILOR trialists. Erlotinib versus docetaxel as second-line treatment of patients with advanced non-small-cell lung cancer and wild-type EGFR tumours (TAILOR): a randomised controlled trial. Lancet Oncol. 2013 Sep;14(10):981-8. doi: 10.1016/S1470-2045(13)70310-3. Epub 2013 Jul 22. PMID 23883922
- [Background] Bouchet F, Geworski L, Knoop BO, Ferrer L, Barriolo-Riedinger A, Millardet C, Fourcade M, Martineau A, Belly-Poinsignon A, Djoumessi F, Tendero K, Keros L, Montoya F, Mesleard C, Martin AL, Lacoeuille F, Couturier O. Calibration test of PET scanners in a multi-centre clinical trial on breast cancer therapy monitoring using 18F-FLT. PLoS One. 2013;8(3):e58152. doi: 10.1371/journal.pone.0058152. Epub 2013 Mar 13. PMID 23516443
- [Background] Laffon E, Bardies M, Barbet J, Marthan R. Calculating an estimate of tissue integrated activity in 18F-FDG PET imaging using one SUV value. EJNMMI Res. 2013 Apr 5;3(1):26. doi: 10.1186/2191-219X-3-26. PMID 23561423
- [Background] Kahraman D, Scheffler M, Zander T, Nogova L, Lammertsma AA, Boellaard R, Neumaier B, Ullrich RT, Holstein A, Dietlein M, Wolf J, Kobe C. Quantitative analysis of response to treatment with erlotinib in advanced non-small cell lung cancer using 18F-FDG and 3'-deoxy-3'-18F-fluorothymidine PET. J Nucl Med. 2011 Dec;52(12):1871-7. doi: 10.2967/jnumed.111.094458. Epub 2011 Nov 7. PMID 22065872